CLINICAL TRIAL: NCT05883475
Title: Investigation of Upper Extremity Function, Sleep Quality, and Functional Independence in Patients With Hemiplegic Shoulder Pain
Brief Title: Effects of Hemiplegic Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 963
Record Dates: First submitted 2023-05-16; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Shoulder Pain
MeSH Terms: conditions — Stroke; Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with shoulder pain: Those who scored above "0" for shoulder pain on the Visual Analog Scale (VAS) were assigned to the group with shoulder pain
  Interventions: Other: Disabilities of the Arm, Shoulder, and Hand Questionnaire; Other: Arm Motor Ability Test; Other: Nine Hole Peg Test; Other: Pittsburg Sleep Quality Index; Other: Functional Independence Measure
- Patients without shoulder pain: Those who scored "0" for shoulder pain on the Visual Analog Scale (VAS) were assigned to the group without shoulder pain
  Interventions: Other: Disabilities of the Arm, Shoulder, and Hand Questionnaire; Other: Arm Motor Ability Test; Other: Nine Hole Peg Test; Other: Pittsburg Sleep Quality Index; Other: Functional Independence Measure

INTERVENTIONS:
Other: Disabilities of the Arm, Shoulder, and Hand Questionnaire — Upper limb function was assessed with the Turkish version of the Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH). The questionnaire DASH is a self-report instrument with 30 items. The total score ranges from 0 to 100, with higher scores indicating a worse upper limb function.
Other: Arm Motor Ability Test — The test assesses hemiparetic upper extremity functional tasks.The increase in the scores of both subparameters of the scale, which is composed of the parameters of functional ability and quality of movement, indicates an improvement in the motor functions of the upper limbs.
Other: Nine Hole Peg Test — Fine motor skills of the upper extremities were assessed.The patient was asked to insert the nine sticks in the box on the table into the holes in the other box as quickly as possible and then remove them immediately. As time increases, fine motor skills of the upper extremities decrease
Other: Pittsburg Sleep Quality Index — Sleep quality was assessed using the this test.This scale, which provides a quantitative measure of sleep quality, is a 19-item self-report scale. The total score greater than 5 indicates "poor sleep quality".
Other: Functional Independence Measure — This test assessed functional capacity in activities of daily living.The higher a person's score, the higher the level of independence.

SUMMARY:
The purposes of this study is to investigate the differences in upper extremity function, sleep quality, and functional independence between patients with and without hemiplegic shoulder pain (HSP).

HSP is defined as musculoskeletal pain in the affected shoulders of individuals after stroke.Numerous studies have found an association between post-stroke shoulder pain and range of motion, sensory impairment, subluxation, spasticity, and complex regional pain syndrome. HSP is a problem that, starting from mild discomfort, leads to gradual functional impairment, ultimately resulting in increasing disability and decreased independence.In the literature, the relationship between HSP and upper extremity function, functional independence, and sleep quality has not been clarified.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Have had a stroke at least three months ago
* Volunteers who can understand or communicate test instructions

Exclusion Criteria:

* Having a history of shoulder surgery
* Having serious shoulder problems before stroke
* Having other neurological conditions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
DASH | one hour
  Upper limb functions was assessed with DASH, AMAT, and Nine Hole Peg Test.The DASH total score ranges from 0 to 100, with higher scores indicating a worse upper limb function.
AMAT | one hour
  The increase in the scores of both subparameters of the AMAT scale, which is composed of the parameters of functional ability and quality of movement, indicates an improvement in the motor functions of the upper limbs.
Nine Hole Peg Test | one hour
  In the Nine hole peg test, fine motor skills of the upper extremities decrease as time goes on.

SECONDARY OUTCOMES:
Sleep Qaulity | one hour
  Sleep quality was assessed using the Pittsburg Sleep Quality Index (PSQI). The total score ranges from 0 to 21, and a total score greater than 5 indicates "poor sleep quality"
Functional Independence | one hour
  The Functional Independence Measure (FIM) assessed functional capacity in activities of daily living. The FIM Consists of 6 parts and analyzes motor and cognitive functions. The higher a person's score, the higher the level of independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)